CLINICAL TRIAL: NCT02164331
Title: A Multimodal Quality Improvement Intervention Using the JNC Guidelines to Promote Control of Patients' BP in Federally Qualified Health Centers
Brief Title: Blood Pressure (BP) Visit Intensification Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kevin Fiscella, MD, MPH, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18HL117801 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-06-16 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JNC guideline training (Experimental): Providers will receive current JNC guideline training for treating patients with uncontrolled hypertension.
  Interventions: Behavioral: JNC guideline training
- Control (No Intervention): Provider patient panels will be assessed for number of uncontrolled hypertensives before receiving the JNC guidelines training. These baseline characteristics will serve as their control conditions.

INTERVENTIONS:
Behavioral: JNC guideline training — Providers will receive a series of trainings on what the JNC guidelines for treating uncontrolled hypertensives are and strategies for meeting those guidelines.
  Arms: JNC guideline training

SUMMARY:
Aim 1: The purpose of the study is to implement the Seventh Joint National Committee on the Diagnosis, Prevention and Treatment of Hypertension (JNC VII) recommendation for monthly visits for hypertensive patients with uncontrolled blood pressure (BP) using a theoretically-informed, empirically grounded, multimodal quality improvement (QI) intervention.

Aim 2: To improve BP control and reduce disparity in BP through implementation of monthly visits.

Aim 3: To assess potential mediators and moderators of the intervention.

DETAILED DESCRIPTION:
This study is a stepped wedged cluster randomized trial designed to improve management of uncontrolled blood pressure among patients in federally qualified health centers through the auspices of the the Clinical Directors Network Practice-Based Research Network (CDN PBRN).

ELIGIBILITY:
Inclusion Criteria:

* Federally Qualified Health Center in the Clinic Directors Network, Practice Champion, Electronic Medical Record System

Exclusion Criteria:

* Clinicians who have been at the practice less than 6 months, Practices planning to change Electronic Medical Record systems within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of office visits | Baseline and aniticipated at 1 year
  Increase patient visit intensification for patients with uncontrolled blood pressure (BP) until the BP is under control.

SECONDARY OUTCOMES:
Reduction in Blood Pressure | Baseline and anticipated at year
  Providers patient panels will be assessed to understand any changes in blood pressure from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Fiscella, MD MPH, Principal Investigator — University of Rochester; Jonathan Tobin, PhD, Principal Investigator — Clinical Directors Network

REFERENCES:
- [Derived] Fiscella K, He H, Sanders M, Cassells A, Carroll JK, Williams SK, Cornell J, Holder T, Khalida C, Tobin JN. Blood Pressure Visit Intensification in Treatment (BP-Visit) Findings: a Pragmatic Stepped Wedge Cluster Randomized Trial. J Gen Intern Med. 2022 Jan;37(1):32-39. doi: 10.1007/s11606-021-07016-9. Epub 2021 Aug 11. PMID 34379277
- [Derived] Fiscella K, Ogedegbe G, He H, Carroll J, Cassells A, Sanders M, Khalida C, D'Orazio B, Tobin JN. Blood Pressure Visit Intensification Study in Treatment: Trial design. Am Heart J. 2015 Dec;170(6):1202-10. doi: 10.1016/j.ahj.2015.08.022. Epub 2015 Sep 12. PMID 26678642